CLINICAL TRIAL: NCT06769867
Title: (Withdrawal) Validation of a Patient-Specific Generative AI-Based Low-Dose Cerebrovascular 3D-DSA Image Reconstruction Method: a Stepwise, Multicenter, Randomized Crossover Trial
Brief Title: (Withdrawal) AI-Based Low-Dose 3D-DSA Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yaowei Bai, MD, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Patient-Specific Generative AI
Record Dates: First submitted 2025-01-02; First posted 2025-01-10 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cerebrovascular Disease
Keywords: Cerebrovascular; AI; 3D-DSA
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PS-3D-DSA (Experimental): undergo a PS-3D-DSA scan
  Interventions: Radiation: PS-3D-DSA
- classic 3D-DSA (Sham Comparator): undergo a classic 3D-DSA scan
  Interventions: Radiation: classic 3D-DSA

INTERVENTIONS:
Radiation: PS-3D-DSA — undergo a PS-3D-DSA scan
  Arms: PS-3D-DSA
Radiation: classic 3D-DSA — undergo a classic 3D-DSA scan
  Arms: classic 3D-DSA

SUMMARY:
If the participants agree to participate in this study, the participants will undergo two scans (classic 3D-DSA and PS-3D-DSA assisted scan) to compare the imaging effects of both. After the procedure, the investigators will record the radiation exposure and collect DSA images.

DETAILED DESCRIPTION:
Although several previous studies have used deep learning methods to reduce 3D-DSA radiation dose, no prospective clinical trial had yet validated the practical application of these models. Herein, the investigators introduce a patient-specific generative AI-based low-dose cerebrovascular 3D-DSA image reconstruction method (PS-3D-DSA) to reconstruct 3D-DSA images from ultra-sparse 2D projection views and a prospective cohort is used to validate its efficacy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Requires 3D-DSA-guided interventional diagnosis or treatment (e.g., cerebral angiography, cerebral artery chemoembolization) and meets operational indications.
3. Can understand the study's purpose, procedures, potential risks, and benefits, and voluntarily signs a written informed consent form.

Exclusion Criteria:

1. Severe heart or lung disease, such as heart failure or chronic obstructive pulmonary disease (COPD).
2. History of high-dose radiation exams or treatments.
3. Known allergies or severe adverse reactions to iodine contrast agents or other relevant medications.
4. Pregnant or breastfeeding women.
5. Severe comorbidities or chronic diseases (e.g., severe diabetes, renal insufficiency).
6. Severe mental illness or cognitive impairment preventing understanding of the study procedures or providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The radiation dose received by patients during interventional procedures when using two scanning protocols (classic 3D-DSA and PS-3D-DSA) | No more than 6 hours
  Using the built-in radiation monitoring function of interventional surgical equipment (DSA system), the radiation dose (AK，air kerma) received by the patient during the procedure is directly measured and recorded. The collected radiation dose data is documented in the patient's medical records and stored in the research database for subsequent analysis and comparative studies.

SECONDARY OUTCOMES:
The image diagnostic capabilities using two scanning protocols (classic 3D-DSA and PS-3D-DSA) | No more than 1 month
  The secondary outcomes focus on evaluating the performance of interventional radiologists using either PS-3D-DSA or classic 3D-DSA for diagnostic tasks, with accuracy as the primary measure. Specifically, the diagnostic results from multiple radiologists will be compared against the gold standard to determine the level of agreement and diagnostic accuracy. This comparison will involve calculating sensitivity, specificity, and overall accuracy. Furthermore, receiver operating characteristic (ROC) curves will be plotted to assess the diagnostic performance and to visually represent the trade-off between sensitivity and specificity for each method.

OTHER OUTCOMES:
Comparison of image quality using two scanning protocols (classic 3D-DSA and PS-3D-DSA) | No more than 1 month
  Algorithmic performance for image quality and interventional radiologists' scoring of image. Specifically, multiple radiologists will provide subjective ratings of image quality, with the best quality rated as 5 and the worst as 1.
  Image Quality (5 points):
  1. point: The smoothness of the video is very poor, with noticeable stuttering in the animation, making it nearly impossible to provide a smooth viewing experience.
  2. points: The smoothness of the video is poor, with a delayed animation, resulting in a less-than-ideal viewing experience.
  3. points: The smoothness of the video is average, the animation is relatively smooth, offering a satisfactory viewing experience.
  4. points: The smoothness of the video is high, with smooth and natural animation, providing an excellent viewing experience.
  5. points: The smoothness of the video is extremely high, with exceptionally smooth animation, providing an outstanding viewing experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Asch CJ, Velthuis BK, Rinkel GJ, Algra A, de Kort GA, Witkamp TD, de Ridder JC, van Nieuwenhuizen KM, de Leeuw FE, Schonewille WJ, de Kort PL, Dippel DW, Raaymakers TW, Hofmeijer J, Wermer MJ, Kerkhoff H, Jellema K, Bronner IM, Remmers MJ, Bienfait HP, Witjes RJ, Greving JP, Klijn CJ; DIAGRAM Investigators. Diagnostic yield and accuracy of CT angiography, MR angiography, and digital subtraction angiography for detection of macrovascular causes of intracerebral haemorrhage: prospective, multicentre cohort study. BMJ. 2015 Nov 9;351:h5762. doi: 10.1136/bmj.h5762. PMID 26553142
- [Background] Irfan M, Malik KM, Ahmad J, Malik G. StrokeNet: An automated approach for segmentation and rupture risk prediction of intracranial aneurysm. Comput Med Imaging Graph. 2023 Sep;108:102271. doi: 10.1016/j.compmedimag.2023.102271. Epub 2023 Jul 22. PMID 37556901